CLINICAL TRIAL: NCT05231018
Title: A Study on the Feasibility and Efficacy of a Telepsychiatric Approach for or COVID19+ Patients, with Particular Attention to Neurocognitive Evaluations and Clinical Questionnaires, Administered Remotely Before and and After Our Treatment Plan.
Brief Title: A Study on a Digital Platform for COVID19+ Patients, Designed to Facilitate Communication and Mental-health Care During and After Hospitalization.
Acronym: DigiCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DigiCOVID
Record Dates: First submitted 2022-01-31; First posted 2022-02-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Mental Health Impairment; Telemedicine
MeSH Terms: conditions — COVID-19 | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psychotherapy (Experimental): The population of interest includes COVID-19 patients previously or currently hospitalized at the Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico, according to inclusion and exclusion criteria.
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — 8-sessions psychotherapy

SUMMARY:
This study presents a digital mental-health protocol designed to offer remote, personalized support to former or current COVID-19 patients.

A total of 100 subjects will be enrolled. Participation is voluntary, and an extended informed-consent form is signed before any evaluation, assessment or voice/video call. Consent forms are collected remotely for those who have been discharged and are currently in remission and in-person for subjects hospitalized in a COVID-19-ward of either pneumology, internal medicine or infectious disease departments.

Efforts will be made to assess all participants who have completed the minimum required intervention activities: for DigiCOVID, minimum required intervention activities include attending psychotherapy sessions at least 4 times. As the main goal of this project is to evaluate the feasibility, acceptability and usability of DigiCOVID, the investigators will conduct an analysis of the following primary outcome measures in all ITT participants:

1. Assessment of completion rate. Based on our previous studies, the investigators expect that ≥80% of participants will complete the battery of online self-reports:
2. Usability ratings obtained post-DigiCOVID via a 7-point Likert-scale questionnaire (mean rating of all responses). This is a brief and embedded post-study questionnaire on program satisfaction, clarity, and perceived benefits. Participants will rate each sentence on the following 7-point Likert scale: 1 = Completely Agree; 2 = Mostly Agree; 3 = Somewhat Agree; 4 = Undecided; 5 = Somewhat Disagree; 6 = Mostly Disagree; 7 = Completely Disagree. Based on our previous studies, the investigators hypothesize exit survey ratings of at least ≥4.5 ±1.5 on the 7-point Likert scale items;
3. Reported side effects (raw score). Based on our previous findings, the investigators expect 0 adverse events due to program use;
4. Overall program completion rate. Based on previous findings, the investigators hypothesize full program completion in ≥70% study participants.

The secondary outcome measures will be collected at baseline and immediately after the treatment for all participants. The investigators designed DigiCOVID to improve mental wellbeing. Therefore, the investigators will measure the impact of the intervention by looking at pre-post changes in the following outcome measures: the General Health Questionnaire (GHQ-12) (Goldberg, 1988) , the Impact of Event Scale-Revised (IES-R) (Weiss & Marmar, 1997), the General Anxiety Disorder-7 (GAD-7) (Robert L Spitzer et al., 2006), the Insomnia Severity Index (ISI) (Morin et al., 2011), and the Patient Health Questionnaire (PHQ-9) (Kroenke et al., 2001). The investigators expect to observe a significant improvement across all these secondary outcome measures in COVID-19 patients. To verify these experimental hypotheses, the investigators will conduct the analysis based on the pre-intervention (baseline) and post-intervention data using parametric and non parametric statistical tests. The criterion for statistical significance is p < 0.05. Results with p < 0.1 will be described as trends.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. A positive COVID-19 test at the moment of enrolment for subjects in the 'patients' group
3. Adequate sensory and motor abilities, without impairments in vision, hearing and handling devices
4. Access to Internet wireless technologies.
5. A good level of Italian in terms of speaking, reading and writing.

Exclusion Criteria:

1. Present of past medical history of schizophrenia, schizoaffective disorder, delusional disorder, bipolar disorder, current substance abuse, all according to the diagnostic and statistical manual fifth edition (DSM-5) (American Psychiatric Association, 2013).
2. With a diagnosis of cognitive impairment and/or dementia (e.g., mild cognitive impairment, Alzheimer's disease, Parkinson's disease);
3. Intellectual disability defined by a total IQ < 70 in Test di Intelligenza Breve (TIB) (Sartori et al., 1997) or Standard Progressive Raven Matrices (John & Raven, 2003)
4. Severe present medical conditions that could interfere with participation.
5. Present or past suicidal ideation or commitment.
6. Significant impairment in the use of digital and technological devices, in questionnaires and test completions, comprehension or with lack of a compliant behavior in the earliest evaluations.
7. Being enrolled in other clinical trials assessing any psychological, or experimental pharmacological treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of completion rate | 2 years
  On the basis of previous studies, ≥80% of participants are expected to complete the battery of online self-reports
Usability ratings obtained post-DigiCOVID via a 7-point Likert-scale questionnaire | 2 years
  General feasibility tested with a brief and embedded post-study questionnaire on program satisfaction, clarity, and perceived benefits
Reported side effects | 2 years
  On the basis of previous findings, zero side effects are expected.
Program completion rate | 2 years
  About 70% of participants are expected to complete the study.

SECONDARY OUTCOMES:
Improvement in mental wellbeing according to the General Health Questionnaire (GHQ-12) (Goldberg, 1988) | 2 years
  Measurements of the impact of the intervention by looking at pre-post changes in the General Health Questionnaire (GHQ-12) (Goldberg, 1988).
Improvement in mental wellbeing according to , the Impact of Event Scale-Revised (IES-R) (Weiss & Marmar, 1997) | 2 years
  Measurements of the impact of the intervention by looking at pre-post changes in the Impact of Event Scale-Revised (IES-R) (Weiss & Marmar, 1997).
Improvement in mental wellbeing according to the General Anxiety Disorder-7 (GAD-7) (Robert L Spitzer et al., 2006) | 2 years
  Measurements of the impact of the intervention by looking at pre-post changes in the the General Anxiety Disorder-7 (GAD-7) (Robert L Spitzer et al., 2006).
Improvement in mental wellbeing according to the Insomnia Severity Index (ISI) (Morin et al., 2011) | 2 years
  Measurements of the impact of the intervention by looking at pre-post changes in the the Insomnia Severity Index (ISI) (Morin et al., 2011).
Improvement in mental wellbeing according to the Patient Health Questionnaire (PHQ-9) (Kroenke et al., 2001). | 2 years
  Measurements of the impact of the intervention by looking at pre-post changes in the Patient Health Questionnaire (PHQ-9) (Kroenke et al., 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Brambilla, Principal Investigator — Università degli Studi di Milano, Fondazione Policlinico di Milano
Locations (1):
- Paolo Brambilla, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cantu F, Biagianti B, Lisi I, R Zanier E, Bottino N, Fornoni C, Gallo F, Ginex V, Tombola V, Zito S, Colombo E, Stocchetti N, Brambilla P. Psychotherapeutic and Psychiatric Intervention in Patients With COVID-19 and Their Relatives: Protocol for the DigiCOVID Trial. JMIR Res Protoc. 2022 Nov 16;11(11):e39080. doi: 10.2196/39080. PMID 36228130